CLINICAL TRIAL: NCT04934384
Title: The Role of Prehospital eFAST in Accelerating Time to Diagnostics or Definitive Treatment in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Other Study IDs: PreH-eFAST
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Trauma Splenic; Trauma Abdomen; Liver Injury
Keywords: trauma; liver; spleen
MeSH Terms: conditions — Abdominal Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive prehospital eFAST: Patients with a positive prehospital eFAST, independently from their hemodynamic status or other vital signs
  Interventions: Diagnostic Test: prehospital extended focused assessment sonography for trauma
- Negative or not performed prehospital eFAST: Patients with a positive prehospital eFAST, independently from their hemodynamic status or other vital signs
  Interventions: Diagnostic Test: prehospital extended focused assessment sonography for trauma

INTERVENTIONS:
Diagnostic Test: prehospital extended focused assessment sonography for trauma — Sonographic procedure performed in the prehospital environment aiming at evaluating peritoneal free fluid in trauma patients
  Other Names: eFAST

SUMMARY:
Actual literature has demonstrated that prehospital extended focused assessment sonography for trauma (eFAST) could impact on logistic and treatment decisions such as mode of transportation and choice of hospital destination.

However, there are no data with regard to in-hospital effects of a positive prehospital eFAST.

The main objective of this study was to evaluate the effects of prehospital eFAST driven decisions on in hospital time-to-definitive diagnostics or time-to definitive treatment, whichever came first, in a level 1 trauma center.

The goal is to define if this information could have a role in prioritizing patients' access to care in a population of abdominal trauma patients with A-AIS > 1 and a documented liver or spleen injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to emergency department with a ICD-9-CM diagnosis of traumatic liver or spleen injury (codes 8640x, 8641x, 8650x, 8651x)
* Abdominal AIS ≥ 2
* CT scan or operating theatre admission performed within 180 minutes from ED admission

Exclusion Criteria:

* Death before CT scan or OR/Angio suite admission (missing primary outcome measure)
* Transferred to other hospitals before CT scan or operating room admission
* Missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve all the patients admitted to the Maggiore Hospital's emergency department (ED) from January 2014 to December 2019 with a traumatic liver or spleen injury who survived enough time to get a CT scan or a surgical intervention within 3 hours from the ED admission
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Time to definitive diagnostics or treatment | 180 minutes
  Time from the ED arrival to CT scan imaging or surgical intervention (whichever came first)

SECONDARY OUTCOMES:
Prehospital time | 240 minutes
  Time from EMS dispatch to ED arrival
Sensitivity and specificity of prehospital eFAST | 240 minutes
  Sensitivity and specificity of prehospital eFAST calculated considering ED eFAST as the gold standard measure

CONTACTS AND LOCATIONS:
Locations (1):
- Maggiore Hospital Ospedale Maggiore Carlo Alberto Pizzardi AUSL di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Botker MT, Jacobsen L, Rudolph SS, Knudsen L. The role of point of care ultrasound in prehospital critical care: a systematic review. Scand J Trauma Resusc Emerg Med. 2018 Jun 26;26(1):51. doi: 10.1186/s13049-018-0518-x. PMID 29940990
- [Background] Chang R, Kerby JD, Kalkwarf KJ, Van Belle G, Fox EE, Cotton BA, Cohen MJ, Schreiber MA, Brasel K, Bulger EM, Inaba K, Rizoli S, Podbielski JM, Wade CE, Holcomb JB; PROPPR Study Group. Earlier time to hemostasis is associated with decreased mortality and rate of complications: Results from the Pragmatic Randomized Optimal Platelet and Plasma Ratio trial. J Trauma Acute Care Surg. 2019 Aug;87(2):342-349. doi: 10.1097/TA.0000000000002263. PMID 31349348
- [Background] Clarke JR, Trooskin SZ, Doshi PJ, Greenwald L, Mode CJ. Time to laparotomy for intra-abdominal bleeding from trauma does affect survival for delays up to 90 minutes. J Trauma. 2002 Mar;52(3):420-5. doi: 10.1097/00005373-200203000-00002. PMID 11901314
- [Background] El Zahran T, El Sayed MJ. Prehospital Ultrasound in Trauma: A Review of Current and Potential Future Clinical Applications. J Emerg Trauma Shock. 2018 Jan-Mar;11(1):4-9. doi: 10.4103/JETS.JETS_117_17. PMID 29628662
- [Background] Jorgensen H, Jensen CH, Dirks J. Does prehospital ultrasound improve treatment of the trauma patient? A systematic review. Eur J Emerg Med. 2010 Oct;17(5):249-53. doi: 10.1097/MEJ.0b013e328336adce. PMID 20124905